CLINICAL TRIAL: NCT03584165
Title: A Long-term Follow-up Study to Evaluate the Safety and Efficacy of Retinal Gene Therapy in Subjects With Choroideremia Previously Treated With Adeno-Associated Viral Vector Encoding Rab Escort Protein-1 (AAV2-REP1) and in Subjects With X-Linked Retinitis Pigmentosa Previously Treated With Adeno-Associated Viral Vector Encoding RPGR (AAV8-RPGR) in an Antecedent Study
Brief Title: Long-term Safety and Efficacy Follow-up of BIIB111 for the Treatment of Choroideremia and BIIB112 for the Treatment of X-Linked Retinitis Pigmentosa
Acronym: SOLSTICE
Status: Enrolling by invitation | Phase: Phase 3 | Type: Interventional
Sponsor: NightstaRx Ltd, a Biogen Company (Other)
Responsible Party: Sponsor
Organization: Biogen (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 273CH201; 2017-003104-42 (EudraCT Number)
Record Dates: First submitted 2018-06-29; First posted 2018-07-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Choroideremia; X-Linked Retinitis Pigmentosa
Keywords: NightstaRx; Biogen; NSR-REP1; CHM; Gene Therapy; AAV; REP1; AAV8; RPGR
MeSH Terms: conditions — Choroideremia | interventions — Cotoretigene Toliparvovec

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- BIIB111 (Experimental): Participants previously treated with sub-retinal injection of BIIB111 in antecedent studies 273CH301 (NCT03496012) and 273CH203 (NCT03507686) will be enrolled. Participants previously treated with this same sub-retinal injection (rAAV2-REP1) in antecedent studies 20150371 (NCT02553135), Pro00028599 (NCT02077361), THOR-TUE-01 (NCT02671539), CHM09/01 (NCT01461213) and REGEN2015 (NCT02407678) will also be invited for enrollment. This is a follow-up study, investigational product was administered in the previous study.
  Interventions: Genetic: BIIB111
- BIIB112 (Experimental): Participants previously treated with sub-retinal injection of BIIB112 in the antecedent study 274RP101 (NCT03116113) will be enrolled. This is a follow-up study, investigational product was administered in the previous study.
  Interventions: Genetic: BIIB112
- Untreated (No Intervention): Untreated participants who served as controls in the antecedent study 273CH301 (NCT03496012), investigating treatment with BIIB111, will be enrolled. This is a follow-up study, participants will not be administered study medication nor receive a sham surgery.

INTERVENTIONS:
Genetic: BIIB111 — Administered as specified in the treatment arm.
  Other Names: AAV2-REP1; rAAV2-REP1
  Arms: BIIB111
Genetic: BIIB112 — Administered as specified in the treatment arm.
  Other Names: AAV8-RPGR
  Arms: BIIB112

SUMMARY:
The objective of the study is to evaluate the long-term safety and efficacy of a sub-retinal injection of BIIB111 in participants with Choroideremia (CHM) who have been previously treated with BIIB111 and who have exited an antecedent study; these treated participants will be compared with untreated control participants who have exited the STAR (NCT03496012) study and BIIB112 in participants with X-linked retinitis pigmentosa (XLRP) who have been previously treated with BIIB112 and who have exited an antecedent study.

DETAILED DESCRIPTION:
This study was previously posted by NightstaRx Ltd. In October 2020, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

CHM Participants

a. Have participated in and exited from an interventional study that investigated the safety and efficacy of a sub-retinal injection of BIIB111 for CHM.

XLRP Participants

a. Have received a sub-retinal injection of BIIB112 for XLRP and have exited an antecedent study.

Key Exclusion Criteria:

Participants are not eligible for study participation if they meet the following exclusion criterion.

a. In the opinion of the Investigator and/or the Sponsor, it is not in the participant's best interest to participate in the study.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2018-06-04 (Actual); Primary Completion 2026-06-04 (Estimated); Study Completion 2026-06-04 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to 5 years
Ophthalmic Examination Assessment: Intraocular Pressure (IOP) | Up to 5 years
Ophthalmic Examination Assessment: Abnormal Slit Lamp Examination | Up to 5 years
Ophthalmic Examination Assessment: Lens Opacity Grading | Up to 5 years
Ophthalmic Examination Assessment: Anterior Chamber and Vitreous Inflammation | Up to 5 years
Ophthalmic Examination Assessment: Indirect Ophthalmoscopy | Up to 5 years

SECONDARY OUTCOMES:
Change from Baseline in Best-Corrected Visual Acuity (BCVA) | Up to 5 years
  BCVA will be assessed for both eyes using the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. BCVA is to be reported as number of letters read correctly by the participant using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Percentage of Participants with no Decrease from Baseline in BCVA or a Decrease from Baseline in BCVA of <5 ETDRS Letters in Choroideremia (CHM) Participants | Up to 5 years
  BCVA will be assessed for both eyes using the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. BCVA is to be reported as number of letters read correctly by the participant using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Percentage of Participants with an Increase from Baseline in BCVA of ≥10 ETDRS Letters in CHM Participants | Up to 5 years
  BCVA will be assessed for both eyes using the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. BCVA is to be reported as number of letters read correctly by the participant using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Percentage of Participants with an Increase from Baseline in BCVA of ≥15 ETDRS Letters in CHM Participants | Up to 5 years
  BCVA will be assessed for both eyes using the Early Treatment of Diabetic Retinopathy Study (ETDRS) visual acuity (VA) chart. BCVA test should be performed prior to pupil dilation, and distance refraction should be carried out before BCVA is measured. Initially, letters are read at a distance of 4 meters from the chart. If <20 letters are read at 4 meters, testing at 1 meter should be performed. BCVA is to be reported as number of letters read correctly by the participant using the ETDRS Scale (ranging from 0 to 100 letters) in the study eye. The lower the number of letters read correctly on the eye chart, the worse the vision (or visual acuity). An increase in the number of letters read correctly means that vision has improved.
Assessment of Fundus Autofluorescence (AF) at Each Visit | Up to 5 years
  Fundus Autofluoroscence will be performed on both eyes to assess the change in the area of viable retinal tissue. It will be reported in square millimetres (mm^2).
Assessment of Fundus Photography at Each Visit | Up to 5 years
  Fundus photography will be performed on both eyes following the dilation of the participant's pupils.
Assessment of Spectral Domain Optical Coherence Tomography (SD-OCT) at Each Visit | Up to 5 years
  SD-OCT will be performed on both eyes to assess the foveal changes and other potential anatomic changes. The measurements were taken after dilation of the participant's pupil and would be reported in micrometres (µm).
Assessment of Microperimetry at Each Visit | Up to 5 years
  Microperimetry will be performed on both eyes to assess changes in retinal sensitivity within the macula. It will be reported in decibels (dB).
Change from Baseline in 25-Item Visual Function Questionnaire (VFQ-25) | Up to 5 years
  VFQ-25 questionnaire measures dimensions of self-reported vision-targeted health status that are most important to persons with eye disease. Total score ranges from 0-100, where a score of 0 represents the worst outcome and 100 represents the best outcome.
Change from Baseline in Visual Field | Up to 5 years
  The outcome measure will be assessed in BIIB112-treated participants.
Percentage of Participants with an Increase from Baseline in Luminance Visual Acuity (LLVA) of ≥10 ETDRS Letters in BIIB112-treated Participants | 18 Months to 60 Months, Post-Day 0 Visits
  The LLVA was measured by placing a 2.0-log-unit neutral density filter over the best correction for that eye and having the participant read the normally illuminated ETDRS chart. The assessment was performed prior to dilating the eyes. Initially, letters are read at a distance of 4 metres from the chart. If <20 letters are read at 4 metres, testing at 1 metre should be performed. BCVA is to be reported as number of letters read correctly by the participant.
Percentage of Participants with an Increase from Baseline in Luminance Visual Acuity (LLVA) of ≥15 ETDRS Letters in BIIB112-treated Participants | 18 Months to 60 Months, Post-Day 0 Visits
  The LLVA was measured by placing a 2.0-log-unit neutral density filter over the best correction for that eye and having the participant read the normally illuminated ETDRS chart. The assessment was performed prior to dilating the eyes. Initially, letters are read at a distance of 4 metres from the chart. If <20 letters are read at 4 metres, testing at 1 metre should be performed. BCVA is to be reported as number of letters read correctly by the participant.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (25):
- United States (10):
  - UCLA - Jules Stein Eye Institute, Los Angeles, California
  - Vitreo Retinal Associates PA - The Millennium Center, Gainesville, Florida
  - University of Miami, Miami, Florida
  - Johns Hopkins Hospital, Baltimore, Maryland
  - MEEI Massachusets Eye and Ear Infirmary, Boston, Massachusetts
  - Columbia University Medical Center, New York, New York
  - Cincinnati Eye Institute - Blue Ash, Cincinnati, Ohio
  - OHSU - Casey Eye Institute, Portland, Oregon
  - Retina Foundation of the Southwest, Dallas, Texas
  - University of Wisconsin School of Medicine, Madison, Wisconsin
- Instituto Genetica Ocular, São Paulo, Brazil
- Canada (3):
  - The Northern Alberta Clinical Trials and Research Centre, Edmonton, Alberta
  - The University of British Columbia - Eye Care Centre, Vancouver, British Columbia
  - McGill University Health Centre, Montreal, Quebec
- Rigshospitalet-Glostrup, Oejenafdelingen, Glostrup Municipality, Denmark
- Helsinki University Central Hospital (HUCH), Helsinki, Finland
- France (2):
  - CHU Montpellier - Saint Eloi, Montpellier
  - Centre Hospitalier National d Ophtalmologie (CHNO) des Quinze-Vingts, Paris
- Germany (2):
  - Universitäts-Augenklinik Bonn, Bonn
  - Universitats Klinikum Tubingen - Institute for Ophthalmic Research, Tübingen
- Radboudumc, Nijmegen, Netherlands
- United Kingdom (4):
  - Moorfields Eye Hospital, London
  - Manchester Royal Eye Hopsital, Manchester
  - John Radcliffe Hospital, Oxford
  - Southampton General Hospital, Southampton

IPD SHARING:
Plan to Share IPD: No